CLINICAL TRIAL: NCT01877226
Title: An Open-Label, Sequential Treatment Study to Assess the Single and Multiple Dose Pharmacokinetics of a New Tapentadol Prolonged-Release 250 mg Formulation in Healthy Subjects
Brief Title: Phase 1 Pharmacokinetic Study of Tapentadol Prolonged-Release 250 Milligram (mg) Formulation in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR015466; R331333PAI1036
Record Dates: First submitted 2013-06-11; First posted 2013-06-13 (Estimated); Last update posted 2013-06-13 (Estimated); Status verified 2013-06

CONDITIONS: Healthy
Keywords: Healthy; Tapentadol
MeSH Terms: interventions — Tapentadol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Tapentadol (Experimental): Tapentadol tamper resistant prolonged-release formulation (TRF) will be administered as 250 milligram oral tablet once (in the morning, 30 minutes after breakfast) on Day 1 and 6, and twice daily (in the morning, 30 minutes after breakfast and in the evening) on Day 4 and 5.
  Interventions: Drug: Tapentadol

INTERVENTIONS:
Drug: Tapentadol — Tapentadol tamper resistant prolonged-release formulation (TRF) will be administered as 250 milligram oral tablet once (in the morning, 30 minutes after breakfast) on Day 1 and 6, and twice daily (in the morning, 30 minutes after breakfast and in the evening) on Day 4 and 5.

SUMMARY:
The purpose of this study is to evaluate pharmacokinetics (explores what the body does to the drug), safety and tolerability of single and multiple-dose of tapentadol in healthy participants.

DETAILED DESCRIPTION:
This is an open-label (all people know the identity of the intervention), single-center, Phase 1 and, single and multiple-dose study of tapentadol tamper resistant prolonged-release formulation (TRF) 250 milligram (mg) tablet in healthy participants. The total study duration will be approximately of 29 days per participant. The study consists of 3 parts: Screening (that is, 21 days before study commences on Day 1); Treatment (single-dose of tapentadol on Day 1, and multiple dose from Day 4-6 [followed by washout period of 24 hours]); and End-of-study (Day 8). All the eligible participants will receive single oral dose of tapentadol TRF 250 mg on Day 1 and twice daily from Day 4-6 (total 5 doses). Participants will keep upright position until 4 hours after study drug administration. Study drug will be administered 30 minutes after breakfast in the morning. Blood samples will be collected for evaluation of pharmacokinetics at pre-dose and post-dose of study treatment. Participants' safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Deemed healthy on the basis of pre-study physical examination, medical history, 12-lead electrocardiogram (ECG), vital signs, and clinical laboratory parameters performed within 2 and 21 days before first study drug administration
* Received a thorough explanation of the optional pharmacogenomic research component of the study and was offered an opportunity to participate by signing the separate pharmacogenomic informed consent document
* Female participants must be postmenopausal (at least 12 months since last menses), surgically sterile, or, if of childbearing potential or sexually active, be practicing an effective method of birth control before entry and throughout the study
* Female participants must have a negative serum beta-human chorionic gonadotropin (b-hCG) pregnancy test at Screening
* Body mass index between 20 and 28 kilogram per square meter (kg/m^2), inclusive, and body weight not less than 50 kilogram

Exclusion Criteria:

* Participants with history of seizure disorder or epilepsy mild or moderate traumatic brain injury, stroke, transient ischemic attack, or brain neoplasm within 1 year of Screening, or severe traumatic brain injury
* History of gastrointestinal disease affecting absorption, gastric surgery or history of or current significant medical illness including cardiac arrhythmias (uneven heart beat) or other cardiac disease, hematologic disease, coagulation disorders lipid abnormalities, significant pulmonary disease,diabetes mellitus, renal or hepatic insufficiency, thyroid disease, neurologic or psychiatric (mental disorders) disease, infection, or any other illness that the investigator considers should exclude the participant - History of clinically significant allergies, especially known hypersensitivity or intolerance or contraindications to opioids, opioid antagonists, benzodiazepines, any study drug formulation component, any of the excipients of the formulation, or heparin
* History of, or a reason to believe a participant has a history of lifetime opioid abuse or, drug or alcohol abuse within the past 5 years
* Positive test for drugs of abuse, such as cannabinoids, alcohol, opiates, cocaine, amphetamines, benzodiazepines, or barbiturates at Screening or on Day -1 of the first treatment period

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2008-09; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Maximum Serum Concentration (Cmax) of Tapentadol | Pre-dose, 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 16, 24, 36, 48 hours post-dose of tapentadol on Day 1 and 6, and pre-dose, 4, 12, 16, 24, 28, 36, 40 hours post multiple-dose administration of tapentadol on Day 4
  The Cmax is the maximum plasma concentration.
Time to Reach Maximum Concentration (tmax) of Tapentadol | Pre-dose, 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 16, 24, 36, 48 hours post-dose of tapentadol on Day 1 and 6, and pre-dose, 4, 12, 16, 24, 28, 36, 40 hours post multiple-dose administration of tapentadol on Day 4
  The tmax is time to reach the maximum observed serum concentration.
Area Under the Serum Concentration-Time Curve From Time Zero to Last Quantifiable Time (AUC [0-last]) of Tapentadol | Pre-dose, 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 16, 24, 36, 48 hours post-dose of tapentadol on Day 1 and 6, and pre-dose, 4, 12, 16, 24, 28, 36, 40 hours post multiple-dose administration of tapentadol on Day 4
  The AUC (0-last) is the area under the serum concentration-time curve from time zero to last quantifiable time.
Area Under the Serum Concentration-Time Curve From Time Zero to Infinite Time (AUC [0-infinity]) of Tapentadol | Pre-dose, 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 16, 24, 36, 48 hours post-dose of tapentadol on Day 1 and 6, and pre-dose, 4, 12, 16, 24, 28, 36, 40 hours post multiple-dose administration of tapentadol on Day 4
  The AUC (0-infinity) is the area under the serum concentration-time curve from time zero to infinite time, calculated as the sum of AUC(last) and C(last)/lambda(z), wherein AUC(last) is area under the serum concentration-time curve from time zero to last quantifiable time; C(last) is the last observed quantifiable concentration; and lambda(z) is elimination rate constant.
Percentage of AUC (0-infinity) Obtained by Extrapolation | Pre-dose, 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 16, 24, 36, 48 hours post-dose of tapentadol on Day 1 and 6, and pre-dose, 4, 12, 16, 24, 28, 36, 40 hours post multiple-dose administration of tapentadol on Day 4
  Percentage of AUC (0-infinity) will be obtained by extrapolation and calculated as: difference between AUC (0-infinity) and AUC (0-last)/AUC (0-infinity) multiplied by 100.
Elimination Half-Life (t [1/2] Lambda) of Tapentadol | Pre-dose, 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 16, 24, 36, 48 hours post-dose of tapentadol on Day 1 and 6, and pre-dose, 4, 12, 16, 24, 28, 36, 40 hours post multiple-dose administration of tapentadol on Day 4
  Elimination half-life (t [1/2] Lambda) is associated with the terminal slope (lambda [z]) of the semi logarithmic drug concentration-time curve, calculated as 0.693/lambda(z).
Rate Constant (Lambda[z]) | Pre-dose, 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 16, 24, 36, 48 hours post-dose of tapentadol on Day 1 and 6, and pre-dose, 4, 12, 16, 24, 28, 36, 40 hours post multiple-dose administration of tapentadol on Day 4
  Lambda(z) is first-order rate constant associated with the terminal portion of the curve, determined as the negative slope of the terminal log-linear phase of the drug concentration-time curve .
Time (t [last])to Reach Last Quantifiable Serum Concentration | Pre-dose, 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 16, 24, 36, 48 hours post-dose of tapentadol on Day 1 and 6, and pre-dose, 4, 12, 16, 24, 28, 36, 40 hours post multiple-dose administration of tapentadol on Day 4
  The t (last) is the time to last quantifiable serum concentration.
Maximum Steady-State Serum Concentration (Cmax,ss) of Tapentadol | Pre-dose, 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 16, 24, 36, 48 hours post-dose of tapentadol on Day 1 and 6, and pre-dose, 4, 12, 16, 24, 28, 36, 40 hours post multiple-dose administration of tapentadol on Day 4
  The Cmax,ss is the observed maximum serum concentration during a dosing interval at steady-state (time at which serum concentration does not change with time).
Trough Serum Concentration (C trough) | Pre-dose, 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 16, 24, 36, 48 hours post-dose of tapentadol on Day 1 and 6, and pre-dose, 4, 12, 16, 24, 28, 36, 40 hours post multiple-dose administration of tapentadol on Day 4
  The C trough is the trough serum concentration before each dose of the multiple-dose treatment.
Time to Reach Maximum Steady-State Serum Concentration (Tmax,ss) of Tapentadol | Pre-dose, 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 16, 24, 36, 48 hours post-dose of tapentadol on Day 1 and 6, and pre-dose, 4, 12, 16, 24, 28, 36, 40 hours post multiple-dose administration of tapentadol on Day 4
  The Tmax,ss is the time to reach the maximum serum concentration after the fifth dose of the multiple-dose treatment.
Area Under the Serum Concentration-Time Curve From Time Zero to tau (AUC [0-tau]) of Tapentadol | Pre-dose, 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 16, 24, 36, 48 hours post-dose of tapentadol on Day 1 and 6, and pre-dose, 4, 12, 16, 24, 28, 36, 40 hours post multiple-dose administration of tapentadol on Day 4
  The AUC (0-tau) is the area under the serum concentration-time curve during a dosing interval (tau).
Steady-State Average Serum Concentration (Cavg,ss) of Tapentadol | Pre-dose, 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 16, 24, 36, 48 hours post-dose of tapentadol on Day 1 and 6, and pre-dose, 4, 12, 16, 24, 28, 36, 40 hours post multiple-dose administration of tapentadol on Day 4
  The Cavg,ss is the average serum concentration at steady-state, calculated as AUC (tau) divided by tau.
Fluctuation Index (FI) | Pre-dose, 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 16, 24, 36, 48 hours post-dose of tapentadol on Day 1 and 6, and pre-dose, 4, 12, 16, 24, 28, 36, 40 hours post multiple-dose administration of tapentadol on Day 4
  The FI is percentage fluctuation that is, variation between peak and trough at steady-state, calculated as difference between Cmax and Ctrough divided by Cavg,ss and multiplied by 100.
Accumulation Ratio | Pre-dose, 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 16, 24, 36, 48 hours post-dose of tapentadol on Day 1 and 6, and pre-dose, 4, 12, 16, 24, 28, 36, 40 hours post multiple-dose administration of tapentadol on Day 4
  Accumulation Ratio calculated for AUC as AUC (x, ss) divided by AUC (x, sd) and for Cmax as C(max,ss) divided by C(max,sd).

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L.C Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.
Locations (1):
- Utrecht, Netherlands

REFERENCES:
- See also: An open-Label, Sequential Treatment Study to Assess the Single- and Multiple-Dose Pharmacokinetics of a new Tapentadol Extended -Release 25-milligram Formulation in Healthy Subjects — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=2253&filename=CR015466_CSR.pdf